CLINICAL TRIAL: NCT06762353
Title: Supportive Peri-implant Care Frequency After Surgical Treatment of Peri-implantitis - a Multi-center Randomized Clinical Trial
Brief Title: SPIC Frequency After Surgical Treatment of Peri-implantitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Giacomo Baima, Co-Principal Investigator (together with Mario Romandini), University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPIC Multi-center
Record Dates: First submitted 2024-12-09; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3-month frequency of supportive peri-implant care (SPIC) (Experimental): SPIC provided at a 3-month frequency starting from the 1-month re-evaluation after surgical treatment of peri-implantitis.
  Interventions: Procedure: 3-month supportive peri-implant care (SPIC)
- 6-month frequency of supportive peri-implant care (SPIC) (Active Comparator): SPIC provided at a 6-month frequency starting from the 1-month re-evaluation after surgical treatment of peri-implantitis.
  Interventions: Procedure: 6-month supportive peri-implant care (SPIC)

INTERVENTIONS:
Procedure: 3-month supportive peri-implant care (SPIC) — SPIC including update on smoking status, evaluation of the patient's adherence to self-performed oral hygiene procedures, full-mouth supra-gingival instrumentation around teeth, repeated sub-gingival instrumentation on sites presenting a PPD >4 mm with BoP/SoP or a PPD≥6 mm, supra-marginal instrumentation around implants, using an erythritol air abrasive system and interdental brushes, sub-marginal instrumentation on implants with BoP after deep probing by an erythritol air abrasive system and/or ultrasonic scaler provided at a 3-month frequency after surgical treatment of peri-implantitis.
  Arms: 3-month frequency of supportive peri-implant care (SPIC)
Procedure: 6-month supportive peri-implant care (SPIC) — SPIC including update on smoking status, evaluation of the patient's adherence to self-performed oral hygiene procedures, full-mouth supra-gingival instrumentation around teeth, repeated sub-gingival instrumentation on sites presenting a PPD >4 mm with BoP/SoP or a PPD≥6 mm, supra-marginal instrumentation around implants, using an erythritol air abrasive system and interdental brushes, sub-marginal instrumentation on implants with BoP after deep probing by an erythritol air abrasive system and/or ultrasonic scaler provided at a 6-month frequency after surgical treatment of peri-implantitis.
  Arms: 6-month frequency of supportive peri-implant care (SPIC)

SUMMARY:
The leading hypothesis behind this study is that a 3-month frequency of supportive peri-implant care (SPIC) recalls after surgical therapy of implants affected by severe peri-implantitis yields better results when compared to a 6-month frequency. Thus, the primary aim of this randomized clinical trial is to compare 2 different frequencies of SPIC recalls (3 and 6 months) after surgical treatment of severe peri-implantitis in terms of treatment success (absence of implant loss, probing pocket depth (PPD) ≤ 5 mm at all aspects, bleeding on deep probing ≤1 site/implant, no suppuration at all aspects, bone loss <0.5 mm) at early follow-up (1-year) and implant survival at the 5-year examination. Secondarily, this randomized clinical trial aims to assess the effects of the 2 different frequencies over clinical attachment levels around remaining teeth.

ELIGIBILITY:
Any patient aged 18 years or more, who has at least one implant affected by severe peri-implantitis, and able to sign an informed consent form will be potentially eligible for this trial. Severe peri-implantitis will be defined as the presence of a peri-implant probing pocket depth [PPD] ≥ 6 mm in at least 1 site of the implant, bleeding and/or suppuration on deep probing [dBoP and/or dSoP, respectively] and radiographically documented marginal bone loss > 3 mm (Carcuac et al. 2016; Romandini et al. 2022) on implants in function by at least 12-months. In the absence of baseline radiographs, implants had to present a bone level >3 mm (Romandini et al. 2021b).

Patients fulfilling the above-mentioned inclusion criteria will not be included in the study if they appear to be unable to attend the study-related procedures (including the long-term follow-up visits) or if one or more of the following systemic or local exclusion criteria are detected during the enrolment phase.

Systemic primary exclusion criteria:

* systemic diseases (e.g. uncontrolled diabetes mellitus) or chronic use of medications (e.g. corticosteroids, bisphosphonates) likely to influence the outcome of therapy or which contraindicates the study procedures;
* smoking >10 cigarettes;
* pregnant or nursing women.

Local primary exclusion criteria:

* history of peri-implantitis treatment on the eligible implants in the previous 6 months;
* hopeless implants (>80% of bone loss/level).

A secondary inclusion criterion will be applied 1-month after surgery:

- absence of peri-implant abscess on the implants to be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2031-09-15 (Estimated); Study Completion 2031-09-15 (Estimated)

PRIMARY OUTCOMES:
Treatment success - criterion 1 (yes/no) | 1 year
  Absence of implant loss, probing pocket depth ≤ 5 mm at all aspects, deep bleeding/suppuration on probing ≤1 site/implant, bone loss <0.5 mm
Implant loss (yes/no) | 5 years
  Implant removed, or mobile, or radiographic evidence of complete loss of osseointegration.

SECONDARY OUTCOMES:
Implant loss (yes/no) | 1 and 3 years
  Implant removed, or mobile, or radiographic evidence of complete loss of osseointegration.
Treatment success - criterion 1 | 3 and 5 years
  Absence of implant loss, probing pocket depth ≤ 5 mm at all aspects, deep bleeding/suppuration on probing ≤1 site/implant, bone loss <0.5 mm
Treatment success - criterion 2 (yes/no) | 1, 3, and 5 years
  Absence of: implant loss, bone loss >1 mm and surgical re-treatments.
Plaque presence (yes/no) | 1, 3 and 5 years
  Presence of plaque (binary - presence/absence in at least 1 site)
Plaque extent | 1, 3 and 5 years
  Plaque extent (continuous - number of sites per implant: 0-6 sites)
Probing pocket depth (mm) | 1, 3 and 5 years
  Probing pocket depth (continuous - assessed at the deepest site per implant)
Bleeding on deep probing (yes/no) | 1, 3 and 5 years
  Bleeding on deep probing (binary - presence/absence in at least 1 site)
Soft-tissue level margin (mm) | 1, 3 and 5 years
  Peri-implant soft-tissue margin level from a constant fixed reference point (continuous - greatest implant level increase among the 6 sites)
Keratinised mucosa height (mm) | 1, 3 and 5 years
  Keratinized mucosa height (continuous - midbuccal aspect)
Bleeding on superficial probing | 1, 3 and 5 years
  Bleeding on superficial circumferential probing (categorical - highest implant level value: 0=no sBoP, 1= isolated bleeding spots; 2=confluent red line on margin; 3=heavy or profuse bleeding)
Suppuration (yes/no) | 1, 3 and 5 years
  Suppuration on deep probing (binary - presence/absence in at least 1 site).
Modified Bleeding Index | 1, 3 and 5 years
  Modified Bleeding Index after profound probing (categorical - highest implant level value: 0=no dBoP; 1=isolated bleeding spots; 2=confluent red line on margin; 3=heavy or profuse bleeding)
Radiographic outcomes | 1, 3 and 5 years
  Taking into account the worst site-specific (between mesial and distal) change: bone level change, bone gain >0.5 mm, bone loss >0.5 mm.
Patient- and clinician- esthetic appreciation | Assessed at 1, 3 and 5 years
  Assessment on a 100 mm visual analogue scale (VAS) of both patient- and clinician- esthetic appreciation and overall patient satisfaction.
Total SPIC duration (months) | Assessed at 1, 3 and 5 years
  Total supportive peri-implant care duration in months , number of sub-marginal re-instrumentations at study implants during SPIC appointments, compliance to SPIC regimen, number of surgical retreatments, and rate of adverse events
Number of sub-marginal re-instrumentations at study implants | Assessed at 1, 3 and 5 years
  Number of sub-marginal re-instrumentations at study implants during SPIC appointments
Compliance to SPIC regimen (yes/no) | Assessed at 1, 3 and 5 years
  Compliance to SPIC regimen according to patient randomisation
Number of surgical retreatments | Assessed at 1, 3 and 5 years
  Number of surgical retreatments performed on the study implant during the study time
Rate of adverse events | Assessed at 1, 3 and 5 years
  Rate of adverse events occurred during the study time, both dependent and independent of the study procedures
Full-mouth plaque score (0-100) | 1, 3, and 5 years
  A full-mouth periodontal examination around the remaining dentition (6 sites per tooth/implant) will be performed assessing plaque (presence/absence)
Full-mouth bleeding score (0-100) | 1, 3, and 5 years
  A full-mouth periodontal examination around the remaining dentition (6 sites per tooth/implant) will be performed assessing Bleeding on Probing (presence/absence),
Clinical attachment level around remaining teeth | 1, 3, and 5 years
  Probing pocket depth (PPD) and recession (REC) (negative values when the CEJ is located subgingivally, positive otherwise). Clinical attachment levels (CAL) will be calculated by summing PPD and REC values for each site. Patient-level incidence of clinical attachment loss >2 mm around teeth will be evaluated as a further outcome.
Chairside aMMP-8 assay (positive/negative) | 1, 3, and 5 years
  Chairside active matrix metalloprotease-8 (aMMP-8) assay will be conducted at the study implant site. Positivity will be determined using a threshold value of ≥20 ng/mL.
Molecular analysis in the peri-implant crevicular fluid | 1 month, 6 months, 1, 3 and 5 years
  Cytokines expressed in the peri-implant crevicular fluid will be monitored as additional outcomes to study the mechanistic interplays involved in the potential different clinical response between groups.
Microbiological analysis | 1 month, 6 months, 1, 3, and 5 years
  Shotgun metagenomics will be used to monitor the microbiological profile associated to the clinical condition.

IPD SHARING:
Plan to Share IPD: Undecided